CLINICAL TRIAL: NCT03640221
Title: A Double-blind, Randomized, Parallel 2- Arm Study to Compare the Efficacy of Ertugliflozin Versus Hydrochlorothiazide in Reducing Sympathetic Neural Overactivity in Patients With Hypertension and Recently-diagnosed Type 2 Diabetes Who Are Receiving Background Standard-of-care Cardio-metabolic Therapy With Metformin, an Angiotensin Converting Enzyme Inhibitor or Angiotensin Receptor Blocker, and a Statin.
Brief Title: Ertugliflozin Versus Hydrochlorothiazide in Reducing Sympathetic Neural Overactivity in Patients With Hypertension and Recently-diagnosed Type 2 Diabetes.
Acronym: Ertugliflozin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn prior to IRB approval and enrollment
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 51991
Record Dates: First submitted 2018-08-01; First posted 2018-08-21 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
Keywords: Hypertension; Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ertugliflozin; Sodium-Glucose Transporter 2 Inhibitors; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, parallel 2- arm study, therapy will be randomly allocated 2:1 to Ertugliflozin oral tablet daily (n=20) or hydrochlorothiazide 12.5mg oral tablet (n=10) and followed for three months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Cedars-Sinai Medical Center pharmacy will be responsible for filling individual patient containers, labeling the containers and performing the blinding of the supplies.
  subjects will receive two bottles of either:
  * Ertugliflozin 15mg tablets (active drug) and a placebo for hydrochlorothiazide; or
  * Placebo for ertugliflozin and hydrochlorthiazide 12.5mg capsules (active drug)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): will receive two bottles of Ertugliflozin 15mg tablets (active drug) and a placebo for hydrochlorothiazide.
  Interventions: Drug: Ertugliflozin; Device: Microneurography; Other: SKNA recordings; Other: Static Handgrip; Other: Post-handgrip forearm vascular occlusion; Other: Testing of the Arterial Baroreflex Function
- Active Comparator (Active Comparator): will receive two bottles of Placebo for ertugliflozin and hydrochlorthiazide 12.5mg capsules (active drug)
  Interventions: Drug: Hydrochlorothiazide 12.5mg; Device: Microneurography; Other: SKNA recordings; Other: Static Handgrip; Other: Post-handgrip forearm vascular occlusion; Other: Testing of the Arterial Baroreflex Function

INTERVENTIONS:
Drug: Ertugliflozin — The sodium-glucose cotransporter 2 (SGLT2) inhibitors are an exciting new class of antidiabetic drugs that cause a modest reduction in high blood pressure and large reductions in the risk of cardiovascular disease (CVD) outcomes and renal outcomes in patients with advanced type 2 diabetes and very high CVD risk. However, the mechanistic underpinning of these CVD benefits is not well understood. this arm will allow us to test our hypothesis.
  Other Names: SGLT2 inhibitor
  Arms: Experimental
Drug: Hydrochlorothiazide 12.5mg — comparator arm allow us to mimic the mild anti hypertensive effect seen with the SGLT-2 inhibitors in order to enable us to differentiate whether the cardiovascular protection seen with the SGLT-2 inhibitors is secondary to its antihypertensive effects vs the potential decrease in sympathetics.
  Other Names: mild antihypertensive comparator
  Arms: Active Comparator
Device: Microneurography — Multiunit recordings of postganglionic sympathetic nerve activity will be obtained with unipolar tungsten microelectrodes inserted selectively into skeletal muscle nerve fascicles of the peroneal nerve. The nerve signals are amplified, filtered (bandwidth 700-2000 Hz), rectified and integrated to obtain a mean voltage display of sympathetic nerve activity. Sympathetic bursts are counted by inspection of the neurograms. A deflection on the mean voltage display is counted as a "burst" if it has a minimal signal to noise ratio of 2:1. The interobserver and intraobserver variations in identifying bursts are <10% and < 5%, respectively.
Other: SKNA recordings — SKNA recordings will be captured by placing ECG electrodes on the chest wall. Recordings will be obtained simultaneously with microneurographic recording. The two techniques will undergo identical filtering and processing of the neurophysiologic inputs which are then displayed simultaneously using identical output functions.
Other: Static Handgrip — Subjects will perform static handgrip at 33% MVC for 2 minutes, using a Stoelting recording handgrip dynamometer. Force output will be recorded continuously and displayed on the computer screen in real time to provide the subject with visual feedback. MVC will be determined for each subject at the beginning of each experiment. Subjects will be instructed to avoid straining maneuvers, changes in breathing, and contraction of non-exercising muscles during the experimental protocols. Ratings of perceived exertion (RPE) will be obtained at the end of each exercise by using a 6- to 20-unit Borg scale. Static handgrip at 33% MVC is accompanied by reflex increases in muscle sympathetic nerve activity caused by activation of the acid-sensing unmyelinated muscle afferents.
Other: Post-handgrip forearm vascular occlusion — This will be performed by inflating a pneumatic cuff on the upper exercising arm to suprasystolic pressure (220 mmHg) beginning 10 seconds before the subject stops gripping and ending 2 minutes into the post-exercise period. The vascular occlusion maintains intramuscular acidosis and thus the stimulation of acid-sensing unmyelinated skeletal muscle afferents and their reflex increase in muscle sympathetic nerve activity and BP, while the muscular relaxation eliminates central command and the attendant increase in heart rate (which returns to the baseline level). As soon as the cuff is release and the forearm circulation is restored, muscle sympathetic nerve activity quickly returns to the baseline level and BP soon follows.
Other: Testing of the Arterial Baroreflex Function — We will compare effects of Ertugliflozin vs. low-dose HCTZ on sinoaortic baroreflex function in hypertensive diabetic subjects during both spontaneous fluctuations in arterial pressure and during decreases and increases in arterial pressure induced by the Valsalva maneuver. The aim of this protocol is to determine if the sympathetic nerve, as well as the heart rate, component of the sinoaortic baroreflex can be augmented by the SGLT2 inhibitor. After obtaining stable baseline recordings, arterial pressure, heart rate, and muscle sympathetic nerve activity will recorded during spontaneous fluctuations in BP over 5 minutes and during both decreases in BP during phase III of the Valsavla maneuver and during the phase IV overshoot in BP upon its release. Frequent accurate measurement of arterial pressure will be obtained with a highly-rated oscillometric arm monitor that records 6 BP readings per minute (Welch Allyn Vital Signs Monitor).

SUMMARY:
The sodium-glucose cotransporter 2 (SGLT2) inhibitors are an exciting new class of antidiabetic drugs that cause a modest reduction in high blood pressure and large reductions in the risk of cardiovascular disease (CVD) outcomes and renal outcomes in patients with advanced type 2 diabetes and very high CVD risk. However, the mechanistic underpinning of these CVD benefits is not well understood. Mechanistic studies are needed to define specific biologic targets and thus optimize therapeutic benefits.

Type 2 diabetes mellitus is firmly established as a state of sympathetic neural overactivity, which may contribute to coexistent hypertension, heart failure, sudden cardiac death, macro- and micro-vascular complications of diabetes, and diabetic nephropathy. In patients recently diagnosed with Type 2 diabetes, microelectrode recordings of sympathetic nerve activity (SNA) targeted to the skeletal muscle circulation have shown both:

1. abnormally high resting (ambient) levels of sympathetic nerve activity; and
2. greatly exaggerated increases in sympathetic nerve activity during isometric (static) handgrip exercise.

The purpose of the proposed study is to determine if Ertugliflozin, a SGLT2 inhibitor, constitutes an effective countermeasure against sympathetic overactivity in patients with diagnosed hypertension and recently diagnosed type 2 diabetes by normalizing the high resting level of muscle sympathetic nerve activity (SNA) as measured by intraneural microelectrodes in the peroneal nerve.

Thus, an effective countermeasure is an urgent unmet medical need. The SGLT2 inhibitors hold exciting promise to address this need.

DETAILED DESCRIPTION:
Static handgrip provides unique mechanistic insights into putative therapeutic targets (in this case the SGLT2 inhibitors) within the human autonomic nervous system include examining the reflexes within the nervous system and its response as a result. Static handgrip will require that patients lay down and with the use of a dyanometer (handgrip device which measures the force output generated from the handgrip exercise) and they will squeeze to the maximum of their ability for 30 seconds, then have a relaxation period, and grip again.

Typically responses to the nervous system travel via unmyelinated skeletal muscle nerve fibers (afferent signals) and the brain responds via the central motor command (or voluntary motor effort) which is its communication to the body to indicate the perception of effort needed in order to complete the task at hand. This volitional component of exercise- is the main mechanism driving heart rate during static handgrip.

When activated by exercise-induced skeletal muscle acidosis (as with static handgrip), muscle afferents signal the brain of a mismatch between muscle perfusion and metabolic demand and trigger a reflex increase in sympathetic nerve activity to non-exercising skeletal muscles. This raises blood pressure and shunts blood to the metabolically active muscle groups. Also, with voluntary exercise, the activation of brain pathways leading to the engagement of parallel central inhibition of the vagus nerve. The result is an increase in cardiac sympathetic nerve activity but it has an an insignificant effect on muscle sympathetic nerve activity, which is driven almost entirely by direct input from the afferent signals.

Thus, the investigators hypothesize that, in type 2 diabetes, impaired skeletal muscle energetics requires patients to use excessive voluntary motor effort to perform routine static handgrip, resulting in a parallel augmentation in cardiac sympathetic nerve activity. If Ertugliflozin improves skeletal muscle energetics, the same isometric exercise will require less motor effort which should result in smaller increases in cardiac sympathetic nerve activity and heart rate as well as a lower rating of perceived exertion on the Borg scale (an established index of central command).

The proposed work stands to advance several innovative concepts that could change the clinical approach to the early management of type 2 diabetes:

1. The sympathetic nervous system as a novel therapeutic target in the mechanistic underpinning of how SGLT2 inhibitors protect against major CVD.
2. Hyperfunction of unmyelinated autonomic (skeletal muscle) sensory nerves as a putative abnormal indicator of diabetic autonomic cardiovascular neuropathy.
3. Early SGLT2-mediated correction of sympathetic overactivity in patients with type 2 diabetes could favorably alter the natural history of diabetic autonomic neuropathy.

The proposed methodology incorporates several scientific rigors:

1. Direct measurement of sympathetic nerve action potentials in human patients using intraneural microelectrodes. This is the gold standard for studying the regulation of the sympathetic nervous system in patients.
2. This microneurographic technique is highly quantitative and remarkably reproducible when a given subject is studied repeatedly without intervention. The spatial resolution is a major advantage by permitting recording of postganglionic fibers innervating the skeletal muscle circulation without "interfering noise" from surrounding postganglionic fibers innervating the skin and from muscle spindles. The temporal resolution permits calculation of the primary endpoint which relates sympathetic discharge rate to the cardiac cycle, providing the best indicator that sympathetic regulation is altered by an SGLT2 inhibitor.
3. Skin sympathetic nerve activity recorded using standard ECG chest leads. The rationale is that the stellate ganglion gives off parallel sympathetic fibers to the heart and to the skin of the chest wall. Conscious dog studies in Dr. Peng-Shen Chen's lab at Indiana University show > 70% concordance of bursts in simultaneous recordings from the stellate ganglion, the cardiac sympathetics, and the chest wall skin sympathetics; similar data are obtained from standard non-invasive ECG chest leads using appropriate bandpass filtering and amplification. Collaborative translational data on healthy human subjects in my lab at Cedars-Sinai show that Skin sympathetic nerve activity displays characteristic discharge properties of Skin sympathetic nerve activity recorded with our intraneural microelectrodes: large non-pulse synchronous bursts of activity that increase immediately with the onset of static handgrip preceded by clear anticipatory bursts. Thus, Skin sympathetic nerve activity provides in conscious human patients a novel quantitative measurement of the centrally-influenced/baroreceptor-insensitive component of cardiac sympathetic nerve activity. Dr. Chen has shown large bursts of Skin sympathetic nerve activity trigger episodes of ventricular tachycardia (VT) in some VT patients with implanted automatic defibrillators. So, if SGLT2 inhibitors buffer excessive increases in Skin sympathetic nerve activity at rest or during static handgrip in patients with type 2 diabetes, this could potentially protect against one form of catecholamine-induced sudden cardiac death.
4. CleverCaps Pill Dispensing System- this unique electronic pill bottle system incorporates wireless technology and state-of-the-art methodology for quantifying and optimizing medication compliance. The system sends reminders for each scheduled dose of each pill type and tracks opening and closing of the bottles in real time as well as the weight of the remaining pills.
5. Welch Allyn Spot Vital Signs Monitor-- provides vital signs in seconds with hospital-grade technology and received an AA rating for continuous inflation mode which takes 6 readings per inflation sequence. This will allow for close titration of medications to induce a 10mmHg bidirectional changes in the mean arterial pressure.
6. the investigators will conduct careful pharmacologic quantitative testing of the baroreceptor reflex.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetes mellitus established < 24 months before enrollment
2. Ages 30-65 years
3. Men and women, inclusive or race/ethnic groups
4. Background standard-of-care cardiometabolic therapy including a stable dose regimen for 6 weeks of: a) metformin and b) an ACEI or an ARB and c) any statin.
5. HBA1C of 6.5 to 8.0
6. Urine albumin/creatinine < 300
7. eGFR > 60
8. Systolic BP 130 to 150 mmHg on the first screening visit and a Systolic BP of 130 to 145 mmHg on the second screening visit
9. BMI 25 to 35 inclusive
10. Normal sinus rhythm by 12-lead ECG with no major conduction abnormalities
11. Left ventricular ejection fraction > 50% by transthoracic echocardiogram
12. Willing and able to cooperate with all aspects of the protocol;
13. Willing and able to give written informed consent for study participation and provide consent for access to medical data according to appropriate local data protection legislation, allowing authorization to access medical records and describe events captured in the endpoints

Exclusion Criteria:

1. Known history of previous cardiovascular disease (CVD)
2. Currently on other diabetes medications such as: insulin analogs, GLP-1 analogs, DPPIV inhibitors, thiazolidinediones, sulfonylureas, meglitinides, alpha glucosidase inhibitors, amylin analogies.
3. Any concomitant medications or supplements, with the exception of: aspirin, ACE-I or ARB, and statin therapy
4. Diagnosed diabetic peripheral sensory neuropathy or retinopathy
5. Orthostatic hypotension defined as standing BP < 100/60 or postural fall of SBP > 20 or DBP > 10
6. Female patients who are pregnant, intend to become pregnant during the study, or are nursing
7. Known hypersensitivity to SGLT-2 inhibitors
8. Presence of hepatic disease
9. History of diabetic ketoacidosis
10. Type 1 diabetes
11. Pancreas or beta-cell transplantation
12. Pancreatitis or pancreatic surgery
13. Unable to communicate or cooperate with the investigator due to language, poor mental development or impaired cerebral function.
14. History of illicit drug use
15. Any other condition(s) deemed by the physician-investigators to be unsafe to participate

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (bursts/minute) | 3 months
  The primary outcome is the change from baseline in muscle sympathetic nerve activity after 3 months of daily treatment with either Ertugliflozin or hydrochlorothiazide. Muscle sympathetic nerve activity will be measured with microelectrodes inserted into the peroneal nerve (microneurography).

SECONDARY OUTCOMES:
Outcome 2 is the increase in muscle sympathetic nerve activity in bursts/minute induced by static handgrip. | 3 months
  Muscle sympathetic nerve activity will be measured at rest and after 2 minutes of static (isometric) handgrip at 33% maximum voluntary contraction. This exercised-induced response will be measured at baseline and after 3 months of Ertugliflozin or HCTZ.
Increase in muscle sympathetic nerve activity induced by post-hand grip forearm vascular occlusion | 3 months
  Muscle sympathetic nerve activity will be measured at rest and after 2 minutes of by post-handgrip forearm vascular occlusion. After 2 minutes of static handgrip at 33% maximum, a pneumatic cuff will be inflated on the upper exercised arm for 2 minutes. This response will be measured at baseline and after 3 months of Ertugliflozin or HCTZ.
Change in chest wall skin sympathetic nerve activity in bursts per minute. | 3 months
  Chest wall skin sympathetic nerve activity, a non-invasive measure of cardiac sympathetic nerve activity, will be measured from standard surface ECG leads using appropriate filtering and amplification.
Arterial baroreflex gain. | 3 months
  Baroreflex gain will be measured as the reflex increase in muscle sympathetic nerve activity in bursts/minutes per mm Hg peak decrease in mean arterial pressure induced by Valsalva strain (Phase III) and the reflex decrease in muscle sympathetic nerve activity per mm Hg during the peak overshoot in mean arterial pressure upon release of the Valsalva maneuver (Phase IV).

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No